CLINICAL TRIAL: NCT06343740
Title: A Pilot Study: A First Evaluation of a Personalized Training Targeting Low Self-esteem: COMET-Y
Brief Title: First Evaluation of COMET-Y
Acronym: COMET-Y
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Accare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSY-2324-S-0136
Record Dates: First submitted 2024-03-19; First posted 2024-04-03 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: Self Esteem; Quality of Life
Keywords: Adolescents; Self Esteem; Mental Health Problems; Quality of Life; Ecological Momentary Assesment

STUDY DESIGN:
Intervention Model Description: This pilot study is a pre-post study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMET-Y (Experimental): All participants receive COMET-Y.
  Interventions: Behavioral: COMET-Y

INTERVENTIONS:
Behavioral: COMET-Y — Competitive memory training (COMET) is a transdiagnostic intervention first developed for adults and later adapted to be used in children and adolescents. The adapted version for youth consists of 7 sessions in which participants learn to facilitate activation of functional/positive thoughts instead of relying on dysfunctional/negative thoughts by using positive self-verbalizations, imagery, body posture, and music. In addition, they are challenged to reformulate dysfunctional/negative thoughts into more functional/positive thoughts. As an addition to the original COMET protocol, there is a parent session in which parents receive psycho-education about their influence on self-esteem. Parents learn to be a 'co-therapist' and to support practicing at home and improve generalization.

SUMMARY:
The goal of this pilot study is to evaluate COMET-Y in 22 adolescents (11-18 years) with various mental health problems and low self-esteem. The main questions is: Does COMET-Y, parallel to care as usual (CAU), improve self-esteem?

Before and after the training participants fill in questionnaires to measure self-esteem, mental health problems, resilience, quality of life, emotions and individual goals. Some of the outcomes are measured through diary methods. Youth and therapists will be assessed to evaluate feasibility and acceptability of the COMET-Y training.

DETAILED DESCRIPTION:
Low self-esteem plays an important role in various mental health problems, and targeted treatment of self-esteem could potentially enhance the efficacy of existing treatments. Research in adults shows that self-esteem training improves self-esteem and mental health problems, but in adolescents this is still unknown. COMET-Y is a personalized self-esteem training, specifically developed for adolescents.

In this pilot study, 22 adolescents (11-18 years) with various mental health problems and low self-esteem will be included. Participants receive COMET-Y parallel to care as usual (CAU). Before and after the training participants fill in questionnaires to measure self-esteem, mental health problems, resilience, quality of life, emotions and individual goals. Some of the outcomes are measured through diary methods. Feasibility and acceptability of the COMET-Y training will be evaluated with youth and therapists.

ELIGIBILITY:
Inclusion Criteria:

* sufficient mastery of Dutch to complete the measurements
* age between 11 - 18 years
* having self-esteem below average (based on a score =<15 on the Rosenberg Self-esteem Scale; RSES)
* currently receiving care for a mental disorder, for example (but not limited to) anxiety disorder, depression, eating disorder, attention-deficit/hyperactivity disorder, oppositional defiant disorder, or autism spectrum disorder.
* willingness to participate in weekly sessions

Exclusion Criteria:

• As intensive treatment can restrain the feasibility of attending the 7 weekly sessions of COMET-Y and engage in homework assignments, participants who need acute care are excluded (e.g. crisis, acute suicidality, or psychotic episode).

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Self Esteem | Two weeks before COMET-Y and a week after COMET-Y
  Global self esteem measured with the Rosenberg self-esteem scale (RSES). Range: 0-30, higher score means higher self-esteem.

SECONDARY OUTCOMES:
Domain-specific Self Esteem | Two weeks before COMET-Y and a week after COMET-Y
  Domain-specific self esteem measured with the Competentiebelevingsschaal voor adolescenten (CBSA). Range: 5-20 for each subscale, a higher score means more competence for the specific domains.
Mental Health Problems | Two weeks before COMET-Y and a week after COMET-Y
  Mental health problems measured with the Strengths and Difficulties Questionnaire (SDQ). Range total score: 0-40, with a higher score corresponding to more problems.
Quality of life | Two weeks before COMET-Y and a week after COMET-Y
  Several aspects of quality of life measured with the Kidscreen-27. Range: 0-130, a higher score means a higher quality of life.
Affect | Two weeks before COMET-Y and a week after COMET-Y
  Positive and negative affect, measured with the Positive and negative affects schedule. (PANAS-C). Range: 0-100, with a higher score higher affect (positive or negative).
Resilience | Two weeks before COMET-Y and a week after COMET-Y
  Resilience is measured with the Brief Resilience Scale (BRS). Range: 1-5, a higher score indicates more resilience.
Ecological Momentary Assessments - Global self-esteem | Two weeks before and two weeks after COMET-Y
  Global self-esteem: short-version of the Rosenberg Self-esteem Scale, as part of a short questionnaire filled in three times a day by the participants via their mobile phones.
  Range: 0-16, higher score means higher self-esteem.
Ecological Momentary Assesments - Goal Based Outcome (GBO) tool for young people | Two weeks before and two weeks after COMET-Y
  The Goal-Based Outcome (GBO) tool for young people, as part of a short questionnaire filled in three times a day by the participants via their mobile phones.
  Participants fill in three personalized goals, which they rate on a scale from 1-10, where higher scores indicate improved goal progress.
Ecological Momentary Assesments - Domain-specific self-esteem | Two weeks before and two weeks after COMET-Y
  Domain-specific self-esteem: perceived self-esteem related functioning covering the specific domains measured by the Competentiebelevingsschaal voor Adolescenten. Range: 0-60, where higher scores indicate more competence.

CONTACTS AND LOCATIONS:
Locations (1):
- Accare, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will ask permission to share the pseudonymized data for potential future re-analysis, such as in a individual participant meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be requested after publication.
Access Criteria: A pseudonymised dataset and analysed dataset will be archived so that data can be shared or checked later (FAIR data use) if the participants have agreed to that.